CLINICAL TRIAL: NCT00458601
Title: A Phase II Study of CDX-110 With Radiation and Temozolomide in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Phase II Study of Rindopepimut (CDX-110) in Patients With Glioblastoma Multiforme
Acronym: ACT III
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX110-003; CDX110-003
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2016-08

CONDITIONS: Malignant Glioma
Keywords: EGFRvIII vaccinetemozolomidecancer vaccineimmunotherapy
MeSH Terms: conditions — Glioma | interventions — rindopepimut; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CDX-110 with GM-CSF (Experimental)
  Interventions: Drug: CDX-110 with GM-CSF; Drug: Temozolomide

INTERVENTIONS:
Drug: CDX-110 with GM-CSF — Three biweekly intradermal injections over four weeks followed by monthly injections until tumor progression. Each dose will be 0.8 mL containing approximately 500 mcg CDX-110 and 150 mcg GM CSF.
  Other Names: CDX-110 with sargramostim (GM-CSF) (Leukine®)
Drug: Temozolomide — Maintenance temozolomide will begin after completion of the three initial injections of CDX-110 plus GM-CSF. 150 to 200 mg/m2 for 5 days during each 28-day cycle for a minimum of six cycles or a maximum of 12 cycles, intolerance or progression.
  Other Names: Temodar

SUMMARY:
This study is designed to evaluate the clinical activity of CDX-110 vaccination when given with standard of care treatment (maintenance temozolomide therapy). Study treatment will be given until disease progression and patients will be followed for long-term survival information. Efficacy will be measured by the progression-free survival status at 5.5 months from the date of first dose.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed de novo GBM with documented EGFRvIII expression in tumor tissue.
* Gross total resection followed by conventional chemoradiation therapy without progression of disease.

Exclusion Criteria:

* Presence of diffuse leptomeningeal disease or gliomatosis cerebri.
* Systemic corticosteroid therapy > 2 mg of dexamethasone or equivalent (as defined by the investigator) per day at study enrollment.
* Patients who have undergone stereotactic radiosurgery prior to or following surgical resection, or the placement of Gliadel® Wafers.
* Known allergy or hypersensitivity to KLH, GM-CSF or yeast derived products, or a history of anaphylactic reactions to shellfish proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-08; Primary Completion 2010-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival status | 5.5mo

SECONDARY OUTCOMES:
Safety and tolerability characterized by adverse events (term, grade, frequency). | 2 years
Safety and tolerability characterized by physical examinations. | 2 years
Safety and tolerability characterized by hematologic and metabolic panel (including CBC with differential, electrolytes, BUN, Cr, liver associated enzymes). | 2 years
Safety and tolerability characterized by urinalysis. | 2 years
Safety and tolerability characterized by vital signs. | 2 years
Immune response; T-cell response to vaccine. | 2 years
Immune response; antibody response to vaccine. | 2 years
Immune response; HLA typing. | 2 years
Overall survival. | indeterminate

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Celldex Investigational Site, Orange, California
  - Celldex Investigational Site, San Francisco, California
  - Celldex Investigational Site, Stanford, California
  - Celldex Investigational Site, New Haven, Connecticut
  - Celldex Investigational Site, Gainesville, Florida
  - Celldex Investigational Site, Chicago, Illinois
  - Celldex Investigational Site, Evanston, Illinois
  - Celldex Investigational Site, Boston, Massachusetts
  - Celldex Investigational Site, Lansing, Michigan
  - Celldex Investigational Site, Saginaw, Michigan
  - Celldex Investigational Site, Hackensack, New Jersey
  - Celldex Investigational Site, Amherst, New York
  - Celldex Investigational Site, New York, New York
  - Celldex Investigational Site, Durham, North Carolina
  - Celldex Investigational Site, Cincinnati, Ohio
  - Celldex Investigational Site, Cleveland, Ohio
  - Celldex Investigational Site, Orange, Ohio
  - Celldex Investigational Site, West Chester, Ohio
  - Celldex Investigational Site, Westlake, Ohio
  - Celldex Investigational Site, Philadelphia, Pennsylvania
  - Celldex Investigational Site, Houston, Texas
  - Celldex Investigational Site, San Antonio, Texas
  - Celldex Investigational Site, Salt Lake City, Utah
  - Celldex Investigational Site, Charlottesville, Virginia
  - Celldex Investigational Site, Seattle, Washington

REFERENCES:
- [Result] Schuster J, Lai RK, Recht LD, Reardon DA, Paleologos NA, Groves MD, Mrugala MM, Jensen R, Baehring JM, Sloan A, Archer GE, Bigner DD, Cruickshank S, Green JA, Keler T, Davis TA, Heimberger AB, Sampson JH. A phase II, multicenter trial of rindopepimut (CDX-110) in newly diagnosed glioblastoma: the ACT III study. Neuro Oncol. 2015 Jun;17(6):854-61. doi: 10.1093/neuonc/nou348. Epub 2015 Jan 13. PMID 25586468